CLINICAL TRIAL: NCT03379298
Title: Regional and Traffic-related Air Pollutants Are Associated With Consumption of a High Fat Diet Among Adolescents
Brief Title: Children's Health Study Diet and Air Pollution
Acronym: CHS DIET
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Frank Gilliland, Professor, University of Southern California
Other Study IDs: CHS01
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Diet Habit; Pollution; Exposure; Child Obesity
MeSH Terms: conditions — Feeding Behavior; Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is built upon the existing data in the Children's Health Study to examine the longitudinal association between childhood exposure to air pollutants and changes in diet among adolescents.

ELIGIBILITY:
Inclusion Criteria:

* children of 4th and 7th grades were enrolled from 12 Southern California communities

Exclusion Criteria:

* extreme mean caloric intake (>5000 or < 500 kcal/day) or no demographic information

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children from 12 Southern California communities were enrolled into the study in 4th and 7th grades (1993-1994) and were followed annually until high school graduation (1998-2001).
Sampling Method: Non-Probability Sample
Enrollment: 3142 (Actual)
Dates: Start 1994-01-01 (Actual); Primary Completion 2001-12-30 (Actual)

PRIMARY OUTCOMES:
Dietary behavior | one year before visit date
  self-reported food frequency questionnaire data

REFERENCES:
- [Derived] Chen Z, Herting MM, Chatzi L, Belcher BR, Alderete TL, McConnell R, Gilliland FD. Regional and traffic-related air pollutants are associated with higher consumption of fast food and trans fat among adolescents. Am J Clin Nutr. 2019 Jan 1;109(1):99-108. doi: 10.1093/ajcn/nqy232. PMID 30596809